CLINICAL TRIAL: NCT03887598
Title: A Multi-center Study of Differential Diagnosis Breast Nodules by Ultrasound Artificial Intelligence and Ultrasound Elastography
Brief Title: Application of Ultrasound Artificial Intelligence and Elastography in Differential Diagnosis of Breast Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xin-Wu Cui (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Taizhou Hospital (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Macheng People's Hospital (Unknown); Huangshi Central Hospital (Other); Affiliated Hospital of Jiangsu University (Other); The First People's Hospital of Yichang (Unknown); Yichang Second People's Hospital (Other); Xiangyang Central Hospital (Other); The Second Hospital of Anhui Medical University (Other); Anqing People's Hospital (Unknown); Huainan People's Hospital (Unknown); Wenzhou Central Hospital (Other); Xuzhou First People's Hospital (Unknown); The Central Hospital of Lishui City (Other); Huai'an First People's Hospital (Other); WISCO General Hospital (Unknown); First People's Hospital of Jiangxia District, Wuhan City (Unknown); Enshi State Central Hospital (Unknown); Lianyungang Third People's Hospital (Unknown); First People's Hospital of Xianyang (Other)
Responsible Party: Sponsor-Investigator, Xin-Wu Cui, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2019(S073)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: Artificial Intelligence; Ultrasound; Breast nodule; ECI
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- breast nodule: Those with one or more breast nodules, age 18 or older, upcoming FNAB or surgery and signed informed consent.Those without adverse effects on the test or threatening other candidates, such as mental illness, pregnancy, poor ultrasound image quality, history of breast surgery or breast biopsy, simple cystic nodules, calcification, excessive mass or too small, the S-DetectTM system can not identify the boundary of the tumor, the basic information is incomplete.
  Interventions: Device: Ultrasound diagnosis

INTERVENTIONS:
Device: Ultrasound diagnosis — Ultrasound diagnosis of lesions with Samsung S-Detect and ECI technology

SUMMARY:
The application of computer-aided diagnosis (CAD) technology "S-Detect" enables qualitative and quantitative automated analysis of ultrasound images to obtain objective, repeatable and more accurate diagnostic results. The Elastic Contrast Index (ECI) technique, unlike conventional strain-elastic imaging techniques, can evaluate the elastic distribution in the region of interest. The purpose of the study was to evaluate the differential diagnosis value of ultrasound S-Detect technology for benign and malignant breast nodules and evaluate the differential diagnosis consistency of the ultrasound S-Detect technique and the examiner for benign and malignant breast nodules and explore the differential diagnosis value of Samsung ultrasound elastic contrast Index (ECI) technique for benign and malignant breast nodules.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women and the second leading cause of cancer deaths worldwide. Therefore, early detection of breast cancer and timely treatment are of great significance for controlling and reducing breast cancer mortality. Breast ultrasound is an adjunct to extensive use in the detection of breast cancer, but ultrasound is highly technically dependent on the examiner, and the results are greatly influenced by the subjective nature of the examiner, adding unnecessary surgery and puncture, which causes great problems for clinicians and patients.Moreover, the value of conventional ultrasound in the differential diagnosis of breast mass is still limited, and the emergence of new technologies such as artificial intelligence and elastography has improved the accuracy of ultrasound diagnosis to varying degrees.

S-Detect technology is a computer-aided (CAD) system recently developed by Samsung Medical Center for breast ultrasound to assist in morphological analysis based on the Breast Imaging Reporting and Data System (BI-RADS) description and final assessment.This provides a new way to identify the benign and malignant breast nodules.

The E-Breast technique, unlike conventional strain-elastic imaging technology, performs an elastic analysis of the entire two-dimensional image.Moreover, when measuring the elastic ratio, it is only necessary to place a region of interest (ROI) at the nodule.Compared with the average elasticity of the surrounding area, it is more reflective of the elastic ratio of the mass to the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Had breast lesions detected by ultrasound
2. Age 18 or older
3. Upcoming FNAB or surgery
4. Signing informed consent

Exclusion Criteria:

1. Patients who had received a biopsy of breast lesion before the ultrasound examination
2. Can not cooperate with the test operation
3. Patients who were pregnant or lactating
4. Patients who were undergoing neoadjuvant treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on gender
Study Population: Patients with breast nodules in large tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-01-18 (Estimated); Study Completion 2020-02-18 (Estimated)

PRIMARY OUTCOMES:
Benign or malignant lesions as determined by pathology | Before surgery or biopsy
  The pathological diagnosis of benign or malignant lesions from surgery samples
Elastic ratio | Before surgery or biopsy
  Clear ECI value

CONTACTS AND LOCATIONS:
Overall Officials: Xin-Wu Cui, PhD,MD, Study Chair — Tongji Hospital; You-Bin Deng, PhD,MD, Study Chair — Tongji Hospital
Locations (1):
- Xin-Wu Cui, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not public because of the personal information of the participants

REFERENCES:
- [Result] Choi JH, Kang BJ, Baek JE, Lee HS, Kim SH. Application of computer-aided diagnosis in breast ultrasound interpretation: improvements in diagnostic performance according to reader experience. Ultrasonography. 2018 Jul;37(3):217-225. doi: 10.14366/usg.17046. Epub 2017 Aug 14. PMID 28992680
- [Result] Kowal M, Filipczuk P, Obuchowicz A, Korbicz J, Monczak R. Computer-aided diagnosis of breast cancer based on fine needle biopsy microscopic images. Comput Biol Med. 2013 Oct;43(10):1563-72. doi: 10.1016/j.compbiomed.2013.08.003. Epub 2013 Aug 19. PMID 24034748
- [Result] Di Segni M, de Soccio V, Cantisani V, Bonito G, Rubini A, Di Segni G, Lamorte S, Magri V, De Vito C, Migliara G, Bartolotta TV, Metere A, Giacomelli L, de Felice C, D'Ambrosio F. Automated classification of focal breast lesions according to S-detect: validation and role as a clinical and teaching tool. J Ultrasound. 2018 Jun;21(2):105-118. doi: 10.1007/s40477-018-0297-2. Epub 2018 Apr 21. PMID 29681007
- [Result] Kim K, Song MK, Kim EK, Yoon JH. Clinical application of S-Detect to breast masses on ultrasonography: a study evaluating the diagnostic performance and agreement with a dedicated breast radiologist. Ultrasonography. 2017 Jan;36(1):3-9. doi: 10.14366/usg.16012. Epub 2016 Apr 14. PMID 27184656
- [Derived] Wei Q, Yan YJ, Wu GG, Ye XR, Jiang F, Liu J, Wang G, Wang Y, Song J, Pan ZP, Hu JH, Jin CY, Wang X, Dietrich CF, Cui XW. The diagnostic performance of ultrasound computer-aided diagnosis system for distinguishing breast masses: a prospective multicenter study. Eur Radiol. 2022 Jun;32(6):4046-4055. doi: 10.1007/s00330-021-08452-1. Epub 2022 Jan 23. PMID 35066633